CLINICAL TRIAL: NCT06113926
Title: Racial Discrimination, Pain, and the Buffering Influences of Acknowledgment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Psi Chi (Other); Society for the Psychological Study of Social Issues (Unknown); D.C. Psychological Association (Unknown)
Responsible Party: Principal Investigator, Katarina AuBuchon, PhD Candidate, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 224125
Record Dates: First submitted 2023-10-23; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Pain, Acute
Keywords: discrimination; racism
MeSH Terms: conditions — Acute Pain; Racism

STUDY DESIGN:
Intervention Model Description: Three independent groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exclusion by White "Players" (No Intervention): Excluded by White "players" in an online ball-tossing game (Cyberball).
- Inclusion by White "Players" (No Intervention): Included by White "players" in an online ball-tossing game (Cyberball).
- Exclusion by White "Players" with Bystander Acknowledgment (Experimental): Excluded by White "players" in an online ball-tossing game (Cyberball) with a White bystander acknowledging the exclusion.
  Interventions: Other: Bystander Acknowledgment

INTERVENTIONS:
Other: Bystander Acknowledgment — The experimenter said "That is so messed up that they excluded you in the task. And honestly, I would say it was racist…" acknowledgment of the participants experience, "…this shouldn't have happened, and I'm really sorry it did…" an apology, and "…I'm going to talk to the primary investigators of the study to figure out how we can make sure that this won't happen to other people" a plan of action.
  Arms: Exclusion by White "Players" with Bystander Acknowledgment

SUMMARY:
Black young adults (aged 18-30; N = 92) were racially included (i.e., received the ball an equal number of times) or excluded (i.e., received the ball only once) by other White players in a ball-tossing computer game called Cyberball; White experimenters acknowledged the exclusion for half of the excluded participants. Participants completed a cold-pressor task twice to measure pain sensitivity (threshold, tolerance, and unpleasantness): immediately prior, and after the Cyberball (and acknowledgment) manipulation. Participants also completed a post-manipulation survey examining the psychological effects of racial exclusion and acknowledgment (i.e., psychological needs satisfaction, negative affect, control).

ELIGIBILITY:
Inclusion Criteria:

* Participants identify as Black/African American
* Age 18-30

Exclusion Criteria:

* Past 30-day persistent pain
* Cardiovascular or circulatory disorders
* Diabetes
* Current pregnancy
* Open sores/frostbite on nondominant hand

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Pain Threshold measured with a cold pressor task | Measured immediately after the manipulation (within minutes).
  Time (in seconds) from the participant places their hand in cold water, to telling the experimenter they are experiencing pain.
Pain Tolerance | Measured immediately after the manipulation (within minutes).
  Time (in seconds) from the participant places their hand in cold water, to when they remove their hand from the water.
Pain unpleasantness | Measured immediately after the manipulation (within minutes).
  Measured with a the McGill-Pain Questionnaire Short Form, the degree of unpleasantness the participant reports from the pain.

SECONDARY OUTCOMES:
Psychological Needs Satisfaction; Self Control subscale | Measured immediately after the manipulation (within minutes).
  Needs-Satisfaction Scale (Zadro et al., 2004)
Psychological Needs Satisfaction; Belongingness subscale | Measured immediately after the manipulation (within minutes).
  Needs-Satisfaction Scale (Zadro et al., 2004)
Psychological Needs Satisfaction; Meaningful Existence subscale | Measured immediately after the manipulation (within minutes).
  Needs-Satisfaction Scale (Zadro et al., 2004)
Psychological Needs Satisfaction; Self esteem subscale | Measured immediately after the manipulation (within minutes).
  Needs-Satisfaction Scale (Zadro et al., 2004)

CONTACTS AND LOCATIONS:
Locations (1):
- The George Washington University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Shared data will be available on OSF

REFERENCES:
- [Derived] AuBuchon KE, Stock ML, Mathur VA, Attey B, Bowleg L. Bystander Acknowledgment Mitigates the Psychological and Physiological Pain of Racial Discrimination for Black Young Adults: A Randomized Controlled Trial. J Pain. 2024 Sep;25(9):104560. doi: 10.1016/j.jpain.2024.104560. Epub 2024 May 11. PMID 38735424
- See also: OSF Preregistration — https://doi.org/10.17605/OSF.IO/2QPV8